CLINICAL TRIAL: NCT06026007
Title: Efficacy of Acupressure Versus Traditional Treatment on Reducing Ankle Edema During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Noha Ahmed Fouad Abd-Elrahman, lecturer for physical therapy for women health, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/12/003363
Record Dates: First submitted 2022-07-30; First posted 2023-09-06 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Gestational Edema
Keywords: Edema Leg
MeSH Terms: interventions — Counseling; Acupressure

STUDY DESIGN:
Intervention Model Description: Sixty pregnant women aged 25 to 35 years old and body mass index was ≥ 30 kg/m², will participate in this study. They will be assigned into three equal groups, Group A will receive only traditional physical therapy protocol in the form of advice including elevation, wearing supportive stocking, and avoiding standing in one position for extended periods, and Group B will receive the same traditional treatment as group A in addition to circulatory exercises, 3times per week for 4 weeks; while Group C will receive the same conventional physical therapy protocol in addition to foot acupressure 3times per week for 4 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): patient in this group received advice only for edema relief
  Interventions: Other: advices
- Circulatory exercise group (Experimental): patient in this group received advice in addition to circulatory exercise for edema relief
  Interventions: Other: advices; Other: Traditional physical therapy
- Acupressure group (Experimental): patient in this group received advice in addition to acupressure for edema relief
  Interventions: Other: advices; Other: Acupressure

INTERVENTIONS:
Other: advices — each pregnant woman was advices how to elevate her legs and daily positions to elevate edema
  Other Names: daily advices
Other: Traditional physical therapy — each pregnant woman was advised about daily routine in addition to circulatory exercise
  Other Names: circulatory exercise
  Arms: Circulatory exercise group
Other: Acupressure — each pregnant woman was advised about daily routine in addition to acupressure therapy
  Other Names: acupressure therapy
  Arms: Acupressure group

SUMMARY:
Incidence of ankle edema is high during pregnancy, If left untreated, it may lead to difficulty walking; stiffness; stretched skin which can become itchy and uncomfortable. Acupressure promotes the condition of the circulatory and lymphatic system leading to the elimination of edema. The aim of this study is to investigate the efficacy of acupressure versus traditional physical therapy treatment on ankle edema during pregnancy.

DETAILED DESCRIPTION:
Sixty pregnant women aged 25 to 35 years old and body mass index was ≥ 30 kg/m², will participate in this study. They will be assigned into three equal groups, Group A will receive only traditional physical therapy protocol in the form of advice including elevation, wearing supportive stocking, and avoiding standing in one position for extended periods, and Group B will receive the same traditional treatment as group A in addition to circulatory exercises, 3times per week for 4 weeks; while Group C will receive the same conventional physical therapy protocol in addition to foot acupressure 3times per week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women in their third trimester,
* age ranged from 25-35 years and
* BMI was ≥30Kg/m2.

Exclusion Criteria:

* Pregnant women with skin diseases
* irremovable bracelet,
* decreased functional active range of motion in the affected lower extremity
* any mental or physical disorders.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-05-08 (Actual)

PRIMARY OUTCOMES:
change in foot and ankle edema during pregnancy | Before starting study and after four weeks of intervention
  Foot Volumeter was used to assess foot and ankle edema

SECONDARY OUTCOMES:
level of swelling | Before starting study and after 4 weeks of intervention
  Patient reported oedema Questionnaire was used to determine the level of swelling

CONTACTS AND LOCATIONS:
Overall Officials: noha abd el rhaman, doctoral, Principal Investigator — BUC
Locations (1):
- faculty of physical therapy Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
only data of the study will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will become available after publication
Access Criteria: data will become available after publication